CLINICAL TRIAL: NCT00001188
Title: The Role of Multi-Modality Therapy for the Treatment of High-Grade Soft Tissue Sarcomas of the Extremities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 830212; 83-C-0212
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-11

CONDITIONS: Sarcoma
Keywords: Chemotherapy; Radiation Therapy; Sarcoma; Surgery
MeSH Terms: conditions — Sarcoma

INTERVENTIONS:
Procedure: radiation therapy following surgery

SUMMARY:
Patients with Grade II and III soft tissue sarcomas of the extremity will be randomized to either receive or not receive radiation therapy following surgery for the removal of the local tumor. All patients in this protocol will receive adjuvant chemotherapy.

DETAILED DESCRIPTION:
Patients with Grade II and III soft tissue sarcomas of the extremity will be randomized to either receive or not receive radiation therapy following surgery for the removal of the local tumor. All patients in this protocol will receive adjuvant chemotherapy.

ELIGIBILITY:
Patients must have biopsy-proven soft tissue sarcoma with one of the following diagnoses:

Liposarcoma (round cell or pleomorphic).

Fibrosarcoma.

Malignant fibrous histiocytoma.

Inflammatory malignant fibrous histiocytoma.

Myxoid malignant fibrous histiocytoma.

Malignant giant cell tumor.

Angiomatoid malignant fibrous histiocytoma.

Leiomyosarcoma.

Malignant hemangiopericytoma.

Rhabdomyosarcoma (embryonal, alveolar, pleomorphic or combined).

Soft tissue sarcoma resembling Ewing's sarcoma.

Synovial cell sarcoma.

Epithelioid sarcoma.

Clear cell sarcoma.

Neurofibrosarcoma.

Epithelioid schwannoma.

Malignant triton tumor.

Angiosarcoma.

Mixed malignant mesenchymoma.

Alvelar soft part sarcoma.

Malignant granular cell tumor.

All lesions must be Grade II or III. No patients with Grade I lesions will be acceptable.

Patients must have undergone a limb-sparing procedure in which all gross tumor has been removed.

Clinical evaluation must reveal no evidence of metastatic disease either in regional lymph nodes or more distant sites.

The soft tissue sarcoma must be on the extremity either at or distal to the shoulder joint or at or distal to the hip joint.

The definitive surgical procedure for a primary lesion or for a recurrence must have been performed no longer than four months from the date of randomization.

Patients must not have received any prior chemotherapy or radiotherapy for their sarcoma.

Patients without a history of any other malignant disease except basal cell carcinoma.

Patients who have not had a serious infection, active bleeding disorders, or concomitant severe disease such as cirrhosis, ischemic heart disease, or evidence of severe impairment of renal function.

Patients must be above the age of 30 and do not have a diagnosis of embryonal rhabdomyosarcoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1983-12; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Suit HD, Russell WO, Martin RG. Sarcoma of soft tissue: clinical and histopathologic parameters and response to treatment. Cancer. 1975 May;35(5):1478-83. doi: 10.1002/1097-0142(197505)35:53.0.co;2-1. PMID 1122498
- [Background] Lindberg RD, Martin RG, Romsdahl MM, Barkley HT Jr. Conservative surgery and postoperative radiotherapy in 300 adults with soft-tissue sarcomas. Cancer. 1981 May 15;47(10):2391-7. doi: 10.1002/1097-0142(19810515)47:103.0.co;2-b. PMID 7272893
- [Background] McNeer GP, Cantin J, Chu F, Nickson JJ. Effectiveness of radiation therapy in the management of sarcoma of the soft somatic tissues. Cancer. 1968 Aug;22(2):391-7. doi: 10.1002/1097-0142(196808)22:23.0.co;2-q. No abstract available. PMID 4298242